CLINICAL TRIAL: NCT02524938
Title: PoGlyDRI - Impact of Dietary Polyphenols on Protein Glycation in Type 2 Diabetes Mellitus Subjects With Chronic Renal Insufficiency
Brief Title: Dietary Polyphenols and Glycation in Renal Insufficiency
Acronym: PoGlyDRI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit due to human resourcing
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GN15DI242
Record Dates: First submitted 2015-07-14; First posted 2015-08-17 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic
Keywords: Dietary polyphenols; Protein glycation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Chlorogenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Chlorogenic Acid (CGA) 400mg/day (CGA-enriched coffee)
  Interventions: Dietary Supplement: Chlorogenic Acid (CGA) enriched coffee
- Control group (Sham Comparator): Conventional coffee (habitual diet)
  Interventions: Dietary Supplement: Conventional coffee

INTERVENTIONS:
Dietary Supplement: Chlorogenic Acid (CGA) enriched coffee — Chlorogenic Acid (CGA) enriched coffee Phase I: CGA-enriched coffee provided with a CGA content of 70-90 mg/100g. Daily CGA intake of 400mg.
  Phase II: recommendation for achieving a CGA-rich diet of at least 400mg/day (total polyphenol intake of at least 1g/day)
  Other Names: CGA-enriched diet
  Arms: Treatment group
Dietary Supplement: Conventional coffee — Phase I: conventional coffee provided (low in CGA) Phase II: standard dietary advice
  Other Names: Habitual diet
  Arms: Control group

SUMMARY:
Type 2 diabetes mellitus (T2DM) is associated with an increased risk of kidney failure, with high levels of glycohaemoglobin (HbA1c) presenting a sharper decline in renal function and an increase in the risk of mortality and end-stage renal disease (ESRD). Polyphenols may improve renal insufficiency in patients with diabetes with chlorogenic acids (CGA) one of the principle polyphenol groups in the diet - coffee/tea, stone fruits (especially plums/prunes) and some vegetables (artichoke, chicory). CGA (3-4 cups of coffee) has been associated with 25% lower risk of T2DM and a favourable reduction of HbA1c, blood pressure, and oxidative stress levels. This randomised controlled trial, therefore, aims to evaluate the effect of high CGA food on glycation and oxidative stress in T2DM subjects with early renal insufficiency (glomerular filtration rate of 35-60 mL/min) as well as progression of renal insufficiency and the risk of cardiovascular diseases.

The study will have two phases - phase I, an interventional study of 3 months followed by phase II, an observational study of 21 months.

In phase I, subjects will be randomized into 2 groups: CGA-enriched diet group, or control (habitual) diet group. The treatment group will be provided with a chlorogenic acid-rich food (coffee) with instructions to achieve an intake of 400 mg per day (equivalent to 3-4 coffee cups per day) for 12 weeks. The control group will receive a conventional coffee low in chlorogenic acid.

Participants will attend three sessions during phase I; baseline, 6 weeks, and 12 weeks. At baseline, general information, medical history, dietary habits and medication use will be recorded and a Food Frequency Questionnaire completed. Urine and blood samples will be collected and blood pressure, waist circumference, height and weight recorded. Participants' diet over the previous 3 days will be assessed by estimated food diary analysis.

In phase II, written dietary recommendations will be provided at three time points (months 6, 12 and 24) - treatment group to achieve a CGA-rich diet (total polyphenol intake of at least 1g per day, and at least 400mg per day of CGA) and standard dietary advice for the control group. Anthropometric/dietary data will be collected as well as blood and urine samples to assess markers of renal function, glycation and oxidative stress, and proteomic markers of cardiovascular disease, coronary artery disease and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* type 2 Diabetes Mellitus
* chronic renal insufficiency with persistent eGFR of 35-60mL/min for at least three months
* fluent in English

Exclusion Criteria:

* dialysis therapy (current or previous)
* malignancy
* transplant recipient
* hyperthyroidism
* hypothyroidism
* high dose glucocorticoids (≥250 mg)
* body mass index (BMI) ≥ 45 kg/m2
* special dietary requirements
* take creatine, antioxidants or vitamin supplements
* smoker
* pregnant
* consume >4 cups of tea/coffee per day
* consume >5 portion of fruits and vegetables per day

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Change in glycohaemoglobin (HbA1c) | 3 months
Change in estimated glomerular filtration rate (eGFR) | 21 months

SECONDARY OUTCOMES:
Change in fasting glucose | 3 months
Change in fructosamine | 3 months
Change in advanced glycation end product (AGE) | 3 months
Change in soluble receptor for AGE (sRAGE) | 3 months
Change in F2-isoprostane | 3 months
Change in malondialdehyde (MDA) | 3 months
Change in Urinary Albumin Excretion | 21 months
Change in creatinine | 21 months
Change in blood pressure | 21 months
Change in crystatin C | 21 months
Change in fibrinogen | 21 months
Change in cholesterol | 21 months
Change in C-reactive protein | 21 months
Change in Interleukin-6 | 21 months
Change in thiobarbituric acid reactive substances (TBARS) | 21 months
Change in advanced oxidation protein products (AOPP) | 21 months
Change in 8hydroxy 2'deoxyguanoside (8OhdG) | 21 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Combet, PhD, Principal Investigator — University of Glasgow
Locations (2):
- United Kingdom (2):
  - NHS Greater Glasgow and Clyde, Glasgow
  - University of Glasgow, Glasgow